

August 20, 2019

Sensitivity, specificity, ROC / AUC values were calculated using SPSS software (version 28, IBM). Separate analyses of sensitivity, specificity, ROC / AUC were performed focusing on all lesions, lesions 2 cm in size or greater, and lesions 3 cm in size or greater.